CLINICAL TRIAL: NCT02394548
Title: A Phase I Trial Of Intensity-Modulated Radiation Therapy (IMRT) Using A Contralateral Esophagus Sparing Technique (CEST) In Locally Advanced Non-Small Cell Lung Cancer (NSCLC) And Limited-Stage Small Cell Lung Cancer (LS-SCLC).
Brief Title: Phase I Trial Of IMRT Using A Contralateral Esophagus Sparing Technique (CEST) In Locally Advanced Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Henning Willers, M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-023
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Results first posted 2020-02-24 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Non-small Cell Lung Carcinoma; Small Cell Lung Carcinoma
Keywords: Locally advanced, inoperable non-small cell lung carcinoma; Limited stage small cell lung carcinoma; Acute esophagitis; Intensity-modulated radiation therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Contralateral Esophagus Sparing Technique (CEST) (Experimental): IMRT with CEST and concurrent chemotherapy (any standard-of-care regimen)
  Interventions: Radiation: Contralateral Esophageal Sparing Technique (CEST)

INTERVENTIONS:
Radiation: Contralateral Esophageal Sparing Technique (CEST) — Determine whether CEST decreases rate of severe acute esophagitis

SUMMARY:
This research study is examining the benefit of a novel radiation planning approach on the likelihood of developing severe esophagitis (irritation and inflammation of the esophagus) during the course of radiation therapy with concurrent chemotherapy which is associated with very painful and difficult swallowing.

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational intervention and also tries to define the appropriate dose of the investigational intervention to use for further studies. "Investigational" means that the intervention is being studied.

The U.S. Food and Drug Administration (FDA) has approved radiation with chemotherapy as a treatment option for your disease.

Currently, there are no established rules to avoid esophagitis in the treatment of lung cancer with radiation therapy. We have developed an IMRT-based technique, termed CEST, to reduce the radiation dose to the part of the esophagus that is located opposite to the tumor. The reason behind this approach is that a lower radiation dose causes less esophagus inflammation and irritation and, therefore, may preserve the swallowing function of the esophagus better. In our clinical experience, reducing the radiation dose to part of the esophagus in this fashion has shown the potential to dramatically decrease the likelihood of severe esophagitis in many though not all people with lung cancer. We therefore wish to analyze this technique further.

There is no firm data to indicate that different chemotherapy regimens given at the same time of radiation therapy result in different rates of esophagitis. The Investigators will, therefore, allow any type of standard-of-care chemotherapy regimen at the discretion of the patient's medical oncologist.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet the following criteria on screening examination to be eligible to participate in the study.

* Histologically or cytologically proven diagnosis of NSCLC or SCLC
* NSCLC, patients with clinical stage IIB-IV patients (AJCC, 7th ed.) are eligible, and for SCLC, limited-stage patients are eligible, if documented to be a candidate for definitive radiation and concurrent chemotherapy in the radiation oncologist or medical oncologist clinic note.

  * Stage IV NSCLC patients are eligible only if they have a solitary brain metastasis
  * Patients with non-malignant pleural effusion are eligible. --- If a pleural effusion is present, the following criteria must be met to exclude malignant involvement:

    * When pleural fluid is visible on both the CT scan and on a chest x-ray, a pleuracentesis is required to confirm that the pleural fluid is cytologically negative.
    * Exudative pleural effusions are excluded, regardless of cytology;
    * Effusions that are minimal (ie, not visible on chest x-ray) that are too small to safely tap are eligible.
* Gross tumor (primary tumor or involved lymph node) must be within 1 cm of esophagus on the most recent chest CT scan.
* ECOG performance status 0-1 within 30 days prior to registration;
* Age ≥18
* Women of childbearing potential must indicate that there is not a possibility of being pregnant at the time of enrollment or have a negative serum pregnancy test prior to the initiation of radiation therapy.
* Women of childbearing potential and male participants must practice adequate contraception.
* Patient must provide study-specific informed consent prior to study entry.

Exclusion Criteria:

Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.

* Greater than minimal, exudative, or cytologically positive pleural effusions
* Tumor suspected or known to invade the esophagus
* Prior chemotherapy if this precludes administration of concurrent chemotherapy for protocol treatment. Note that induction chemotherapy is allowed as long as concurrent chemotherapy is possible.
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immuno-compromised patients.
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
* Any history of allergic reaction to chemotherapies used

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-06; Primary Completion 2019-02 (Actual); Study Completion 2021-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henning Willers, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts

REFERENCES:
- [Derived] Kamran SC, Yeap BY, Ulysse CA, Cronin C, Bowes CL, Durgin B, Gainor JF, Khandekar MJ, Tansky JY, Keane FK, Olsen CC, Willers H. Assessment of a Contralateral Esophagus-Sparing Technique in Locally Advanced Lung Cancer Treated With High-Dose Chemoradiation: A Phase 1 Nonrandomized Clinical Trial. JAMA Oncol. 2021 Jun 1;7(6):910-914. doi: 10.1001/jamaoncol.2021.0281. PMID 33830168

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was consented but never began treatment
Period: Overall Study
Arm/Group | Contralateral Esophagus Sparing Technique (CEST)
Started | 26
Completed | 25
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Contralateral Esophagus Sparing Technique (CEST)
Number analyzed (Participants) | 26
Age, Continuous [Median (Full Range); unit: years] | 67 [51 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 3 or Higher Acute Esophagitis (CTCAE)
Description: Esophagitis will be measured using the Common Toxicity Criteria for Adverse Effects (CTCAE) v4 scoring scale
Time Frame: up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Contralateral Esophagus Sparing Technique (CEST)
Number analyzed (Participants) | 26
Participants | 0

2. Secondary Outcome: Number of Participants With Grade 3 or Higher Acute Esophagitis (RTOG)
Description: Esophagitis will be measured using the historical Radiation Therapy Oncology Group (RTOG) scoring scale
Time Frame: Baseline , up to 3 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Contralateral Esophagus Sparing Technique (CEST)
Number analyzed (Participants) | 26
Participants | 0

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events will be measured using CTCAE v4 scoring scale
Time Frame: Baseline, up to 2 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Contralateral Esophagus Sparing Technique (CEST)
Number analyzed (Participants) | 26
Participants | 24

4. Secondary Outcome: Rate of Local and Regional Failure
Description: Response and progression will be evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) guideline. No isolated locoregional tumor failures at a median follow-up of up to 2 years.
Time Frame: Median follow-up of up to 2 years
Measure: Number; unit: locoregional tumor failures
Arm/Group | Contralateral Esophagus Sparing Technique (CEST)
Number analyzed (Participants) | 26
locoregional tumor failures | 0

5. Secondary Outcome: Overall Survival Rate
Description: Follow-up time will be calculated from the date of registration to the date of death or the last follow-up date on which the patient was reported alive. Overall survival rates will be estimated using the Kaplan-Meier method.
Time Frame: 2 Years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Contralateral Esophagus Sparing Technique (CEST)
Number analyzed (Participants) | 26
percentage of participants | 67 [45 to 82]

ADVERSE EVENTS:
Time Frame: From the start of treatment up to 2 years
Description: Serious adverse events were defined as adverse events with a grade of 3 or higher that were deemed to be possibly, probably, or definitely related to treatment.
Arm/Group | Contralateral Esophagus Sparing Technique (CEST)
All-Cause Mortality (participants affected / at risk) | 1/26
Serious Adverse Events (participants affected / at risk) | 21/26
Other Adverse Events (participants affected / at risk) | 18/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Contralateral Esophagus Sparing Technique (CEST) (N=26)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Ventricular Tachycardia (Cardiac disorders) | 1
Hyperglycemia (Blood and lymphatic system disorders) | 1
Heart Failure (Cardiac disorders) | 1
Lymphocyte count decreased (Blood and lymphatic system disorders) | 19
Anemia (Blood and lymphatic system disorders) | 1
Neutrophil count decreased (Blood and lymphatic system disorders) | 11
white blood cell count decreased (Blood and lymphatic system disorders) | 8
Leukocytosis (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Contralateral Esophagus Sparing Technique (CEST) (N=26)
Esophagitis (Respiratory, thoracic and mediastinal disorders) | 8
Fatigue (General disorders) | 6
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Dermatitis Radiation (Skin and subcutaneous tissue disorders) | 5
Erythema (Skin and subcutaneous tissue disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Atrial Fibrillation (Cardiac disorders) | 2
Gerd (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 1
Hyponatremia (Blood and lymphatic system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 3
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Oral Thrush (Gastrointestinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1

LIMITATIONS AND CAVEATS:
This protocol received IRB approval on 7/20/21 to remove secondary outcome "Median Survival Time" so this pre-specified outcome was subsequently deleted from the CT.gov record. The reason is that the secondary outcome of median survival time was not reached at time of analysis and final publication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-22): https://cdn.clinicaltrials.gov/large-docs/48/NCT02394548/Prot_SAP_001.pdf
  • Informed Consent Form (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT02394548/ICF_002.pdf